CLINICAL TRIAL: NCT02207374
Title: Safety and Efficacy of Semaglutide Once Weekly in Monotherapy or in Combination With One OAD in Japanese Subjects With Type 2 Diabetes Who Are Insufficiently Controlled on Diet/Exercise Therapy or OAD Monotherapy
Brief Title: A Trial Comparing the Safety and Efficacy of Semaglutide Once Weekly in Monotherapy or in Combination With One OAD in Japanese Subjects With Type 2 Diabetes
Acronym: SUSTAIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9535-4091; U1111-1140-3081 (Other: WHO); JapicCTI-142640 (Registry Identifier: JAPIC)
Record Dates: First submitted 2014-08-01; First posted 2014-08-04 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Semaglutide 0.5 mg (Experimental)
  Interventions: Drug: semaglutide
- Semaglutide 1.0 mg (Experimental)
  Interventions: Drug: semaglutide
- One additional OAD + pre-trial treatment (Active Comparator): The type and dosage of the additional OAD will be selected by the investigators according to the approved Japanese labelling including drug combinations and contraindications. One of DPP-4 inhibitor (dipeptidyl peptidase-4), SU (sulfonylurea), glinide, biguanide, α-GI (α-glucosidase inhibitor)or TZD (thiazolidinediones) will be selected as the additional OAD. For the subjects treated with OAD monotherapy as pre-trial treatment, the type and dosage of the additional OAD with a different mechanism of action from the pre-trial OAD should be chosen.
  Interventions: Drug: DPP-4 inhibitor

INTERVENTIONS:
Drug: semaglutide — Subject will receive either a dose of 0.5 or 1.0 mg of semaglutide once weekly (subcutaneous (s.c.) injection).Treatment duration 56 weeks.
  Arms: Semaglutide 0.5 mg; Semaglutide 1.0 mg
Drug: DPP-4 inhibitor — Subjects will receive one DPP-4 inhibitor in addition to pre-trial OAD monotherapy, if any, for 56 weeks.
  Arms: One additional OAD + pre-trial treatment

SUMMARY:
This trial is conducted in Asia. The aim of the trial is to investigate safety and efficacy of semaglutide once weekly in monotherapy or in combination with one OAD (oral anti-diabetic drug) in Japanese subjects with type 2 diabetes who are insufficiently controlled on diet/exercise therapy or OAD monotherapy.

All subjects will continue their pre-trial treatment (diet and exercise therapy or OAD monotherapy in addition to diet and exercise therapy) during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at least 20 years at the time of signing informed consent
* HbA1c (glycosylated haemoglobin A1c) between 7.0% and 10.5% (53-91 mmol/mol) (both inclusive)
* Japanese subjects with type 2 diabetes mellitus (diagnosed clinically) and on stable treatment (defined as unchanged medication and unchanged dose) who are: a) on diet and exercise therapy for at least 30 days before Visit 1 (week -2). or b) on OAD monotherapy (either of SU (sulfonylurea), glinide, a-GI (a-glucosidase inhibitor) or TZD (thiazolidinediones)) within approved Japanese labelling in addition to diet and exercise therapy for at least 60 days before Visit 1 (week -2)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using an adequate contraceptive method (e.g., abstinence [not having sex], diaphragm, condom [by the partner], intrauterine device, sponge, spermicide or oral contraceptives) throughout the trial including the 5 week follow-up period
* Treatment with glucose lowering agent(s) other than stated in the inclusion criteria within 60 days before Visit 1 (week -2) and treatment with once weekly glucagon-like peptide-1 (GLP-1) receptor agonists within 90 days before Visit 1 (week -2). An exception is short-term treatment (below or equal to 7 days in total) with insulin in connection with inter-current illness
* Any disorder which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol
* History of chronic or idiopathic acute pancreatitis
* Screening calcitonin value above or equal to 50 ng/L (pg/mL)
* Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2)
* Impaired renal function defined as estimated glomerular filtration rate (eGFR) below 30 mL/min/1.73 m^2 per modification of diet in renal disease (MDRD) formula (4 variable version)
* Acute coronary or cerebrovascular event within 90 days before randomisation (Visit 2 [week 0])
* Heart failure, New York Heart Association (NYHA) class IV

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2016-02-27 (Actual); Study Completion 2016-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (36):
- Japan (36):
  - Novo Nordisk Investigational Site, Akita-shi, Akita
  - Novo Nordisk Investigational Site, Annaka-shi, Gunma
  - Novo Nordisk Investigational Site, Asahikawa-shi, Hokkaido
  - Novo Nordisk Investigational Site, Bunkyo-ku, Tokyo
  - Novo Nordisk Investigational Site, Chuo-ku Tokyo
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Fukuoka
  - Novo Nordisk Investigational Site, Higashiosaka-shi, Osaka
  - Novo Nordisk Investigational Site, Izumisano
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Katsushika-ku, Tokyo
  - Novo Nordisk Investigational Site, Kitakyushu-shi, Fukuoka
  - Novo Nordisk Investigational Site, Koriyama-shi, Fukushima
  - Novo Nordisk Investigational Site, Kumamoto-shi,Kumamoto
  - Novo Nordisk Investigational Site, Kyoto-shi, Kyoto
  - Novo Nordisk Investigational Site, Mito-shi, Ibaraki
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hygo
  - Novo Nordisk Investigational Site, Nishinomiya-shi, Hyogo
  - Novo Nordisk Investigational Site, Okawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Okayama-shi, Okayama
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Oyama-shi, Tochigi
  - Novo Nordisk Investigational Site, Saga-shi,Saga
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Sendai
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Suita-shi, Osaka
  - Novo Nordisk Investigational Site, Takatsuki-shi, Osaka
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Ube-shi, Yamaguchi
  - Novo Nordisk Investigational Site, Yokohama

REFERENCES:
- [Result] Kaku K, Yamada Y, Watada H, Abiko A, Nishida T, Zacho J, Kiyosue A. Safety and efficacy of once-weekly semaglutide vs additional oral antidiabetic drugs in Japanese people with inadequately controlled type 2 diabetes: A randomized trial. Diabetes Obes Metab. 2018 May;20(5):1202-1212. doi: 10.1111/dom.13218. Epub 2018 Feb 21. PMID 29322610
- [Result] Petri KCC, Ingwersen SH, Flint A, Zacho J, Overgaard RV. Exposure-response analysis for evaluation of semaglutide dose levels in type 2 diabetes. Diabetes Obes Metab. 2018 Sep;20(9):2238-2245. doi: 10.1111/dom.13358. Epub 2018 Jun 15. PMID 29748996
- [Result] Carlsson Petri KC, Ingwersen SH, Flint A, Zacho J, Overgaard RV. Semaglutide s.c. Once-Weekly in Type 2 Diabetes: A Population Pharmacokinetic Analysis. Diabetes Ther. 2018 Aug;9(4):1533-1547. doi: 10.1007/s13300-018-0458-5. Epub 2018 Jun 15. PMID 29907893
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 41 sites in Japan.
Pre-assignment Details: Subjects were either on diet and exercise therapy only or on stable treatment on oral anti-diabetic drugs (OADs) mono-therapy [either of sulphonyl urea (SU), glinide, alpha-glucosidase inhibitor (α-GI) or thiazolidinediones (TZD)] within approved Japanese labelling in addition to diet and exercise therapy before week -2.
Groups:
- Semaglutide 0.5 mg: Subjects were randomized to receive semaglutide 0.5 mg once weekly subcutaneously (s.c.; under the skin) in the thigh, abdomen, or upper arm for a period up to 56 weeks. The treatment period was divided into the dose escalation and the dose maintenance period. Subjects followed a fixed dose escalation pattern to mitigate tolerability concerns, starting with once-weekly doses of 0.25 mg for 4 weeks (4 doses), then escalated to once weekly 0.5 mg maintenance dose for 52 weeks (maximum dose). Doses were not changed during the trial after the maintenance dose was reached. Semaglutide 1.34 mg/mL was supplied in a 1.5 mL pre-filled PDS290 pen-injector and administered on the same day of every week during the trial. All subjects continued their pre-trial treatment of either diet and exercise therapy or OAD monotherapy in addition to diet and exercise throughout the trial.
- Semaglutide 1.0 mg: Subjects were randomized to receive semaglutide 1.0 mg once weekly subcutaneously (s.c.; under the skin) in the thigh, abdomen, or upper arm for a period up to 56 weeks. The treatment period was divided into the dose escalation and the dose maintenance period. Subjects followed a fixed dose escalation pattern to mitigate tolerability concerns, starting with once-weekly doses of 0.25 mg for 4 weeks (4 doses), then escalated to once weekly doses of 0.5 mg for 4 weeks, and finally escalated to once weekly 1.0 mg maintenance dose for 48 weeks (maximum dose). Doses were not changed during the trial after the maintenance dose was reached. Semaglutide 1.34 mg/mL was supplied in a 1.5 mL pre-filled PDS290 pen-injector and administered on the same day of every week during the trial. All subjects continued their pre-trial treatment of either diet and exercise therapy or OAD monotherapy in addition to diet and exercise throughout the trial.
- Additional OAD: Subjects were randomised to receive one additional OAD in addition to the pre-trial treatment for a duration of 56 weeks. The type and dosage of the additional OAD was selected by the investigator according to the approved Japanese labelling based on drug combinations and contraindications. One of the following OADs was to be selected as the additional OAD therapy: dipeptidyl peptidase-4 (DPP-4) inhibitor, SU, glinide, biguanide, α-GI and TZD. For subjects treated with OAD as pre-trial treatment, the type and dosage of the additional OAD with a different mechanism of action from the pre-trial OAD was to be chosen. The dose of the additional OAD was optimized within approved Japanese labelling until week 8 (dose adjustment period) and the dose remained unchanged until week 56 (maintenance dose) unless rescue medication was needed. The type of the additional OAD remained unchanged during the trial.
Period: Overall Study
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Additional OAD
Started | 239 | 241 | 121
Exposed | 239 | 241 | 120
Completed | 233 | 231 | 115
Not Completed | 6 | 10 | 6
Not completed — Withdrawal by Subject | 5 | 9 | 4
Not completed — Death | 1 | 0 | 1
Not completed — Missing follow-up information | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects who had received at least one dose of semaglutide 0.5 mg (s.c.), semaglutide 1.0 mg (s.c.) or one additional OAD.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Additional OAD | Total
Number analyzed (Participants) | 239 | 241 | 120 | 600
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (10.6) | 58.7 (10.2) | 59.2 (10.1) | 58.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 67 | 31 | 171
  Male | 166 | 174 | 89 | 429
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.04 (0.89) | 8.14 (0.96) | 8.10 (0.89) | 8.09 (0.92)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AEs) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a product, whether or not considered related to the product. All AEs mentioned here are treatment emergent adverse events (TEAE) defined as an event that had onset date (or increase in severity) on or after the first day of exposure to randomised treatment (week 0-56 treatment period) and no later than the follow-up visit during the on-treatment observation period (date of last dose + 42 days).
Time Frame: Weeks 0-56
Population: The safety analysis set (SAS) included all randomised subjects who had received at least one dose of semaglutide 0.5 mg (s.c.), semaglutide 1.0 mg (s.c.) or one additional OAD. Subjects in the SAS contributed to the evaluation "as treated".
Measure: Number; unit: Number of events
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Additional OAD
Number analyzed (Participants) | 239 | 241 | 120
Number of events | 909 | 954 | 269

2. Secondary Outcome: Number of Severe or Blood Glucose (BG) Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or blood glucose (BG) confirmed symptomatic hypoglycaemic episodes were defined as episodes that were severe and/or BG confirmed by a plasma glucose value of <56 mg/dL (3.1 mmol/L), with symptoms consistent with hypoglycaemia. Severe hypoglycaemia: was an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. The episodes mentioned here are treatment emergent hypoglycaemic episodes and defined as an event that had onset date (or increase in severity) on or after the first day of exposure to randomised treatment (week 0-56 treatment period) and no later than the follow-up visit during the on-treatment observation period (date of last dose + 42 days).
Time Frame: Weeks 0-56
Population: as for outcome 1
Measure: Number; unit: Number of episodes
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Additional OAD
Number analyzed (Participants) | 239 | 241 | 120
Number of episodes | 4 | 8 | 2

3. Secondary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c)
Description: The observed mean change in HbA1c values from baseline after 56 weeks of treatment. Changes in HbA1c were analysed using a mixed model for repeated measurements (MMRM) with treatment and pre-trial treatment at screening as fixed factors and baseline value as covariate. The data were analysed for the "on-treatment without rescue medication" observation period which includes observations noted at or after the date of first dose of randomised treatment and not after the last dose of the trial product (+ a 7-day visit window) or initiation of rescue medication.
Time Frame: Week 0, week 56
Population: The full analysis set (FAS) included all randomised subjects who have received at least one dose of trial product. All subjects contributed to the statistical model of the data analysis, but not all subjects had a value at week 56.
Measure: Least Squares Mean (Standard Error); unit: Percentage (%) of HbA1c
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Additional OAD
Number analyzed (Participants) | 220 | 204 | 106
Percentage (%) of HbA1c | -1.74 (0.05) | -2.03 (0.05) | -0.67 (0.07)

ADVERSE EVENTS:
Time Frame: All AEs mentioned here are treatment emergent adverse events (TEAE), defined as an event that had onset date (or increase in severity) on or after the first day of exposure to randomised treatment (week 0-56 treatment period) and no later than the follow-up visit during the on-treatment observation period (date of last dose + 42 days).
Description: The safety analysis set included all randomised subjects who had received at least one dose of semaglutide 0.5 mg (s.c.), semaglutide 1.0 mg (s.c.) or one additional OAD. Subjects in the SAS contributed to the evaluation "as treated".
Arm/Group | Semaglutide 0.5 mg | Semaglutide 1.0 mg | Additional OAD
Serious Adverse Events (participants affected / at risk) | 19/239 | 12/241 | 8/120
Other Adverse Events (participants affected / at risk) | 160/239 | 169/241 | 61/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=239) | Semaglutide 1.0 mg (N=241) | Additional OAD (N=120)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Drowning (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery angioplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Peripheral revascularisation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peritonsillar abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Varicose vein operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 0.5 mg (N=239) | Semaglutide 1.0 mg (N=241) | Additional OAD (N=120)
Abdominal discomfort (Gastrointestinal disorders) | 15 (15) | 15 (16) | 0 (0)
Amylase increased (Investigations) | 7 (8) | 13 (15) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 13 (13) | 10 (10)
Constipation (Gastrointestinal disorders) | 44 (49) | 36 (40) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 18 (22) | 32 (36) | 0 (0)
Diabetic retinopathy (Eye disorders) | 11 (11) | 16 (16) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 24 (33) | 38 (49) | 8 (9)
Gastroenteritis (Infections and infestations) | 15 (16) | 5 (6) | 2 (2)
Lipase increased (Investigations) | 21 (25) | 33 (36) | 2 (2)
Nasopharyngitis (Infections and infestations) | 81 (132) | 75 (105) | 41 (60)
Nausea (Gastrointestinal disorders) | 29 (38) | 46 (70) | 1 (1)
Pharyngitis (Infections and infestations) | 12 (15) | 9 (9) | 2 (3)
Vomiting (Gastrointestinal disorders) | 13 (17) | 14 (21) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"At the end of the trial, one or more scientific publications may be prepared collaboratively by the Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property".